CLINICAL TRIAL: NCT02339766
Title: Comparison of Intrathecal Morphine With Quadratus Lumborum Block for Post-Cesarean Delivery Analgesia:
Brief Title: Quadratus Lumborum Block for Post-Cesarean Analgesia
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Not feasible due to difficulty with recruitment.
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 106224
Record Dates: First submitted 2015-01-06; First posted 2015-01-15 (Estimated); Last update posted 2021-10-22 (Actual); Status verified 2021-09

CONDITIONS: Postoperative Pain
Keywords: Cesarean; Quadratus Lumborum Block; Analgesia; Ultrasonography
MeSH Terms: conditions — Pain, Postoperative; Agnosia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1 (Sham Comparator): Group 1 will receive intrathecal morphine co-administered with the spinal anesthetic. After the completion of surgery, bilateral ultrasound guided Sham Block be done with 25 mL of saline per side.
  Interventions: Procedure: Sham Block; Drug: Intrathecal Morphine
- Group 2 (Active Comparator): Group 2 will receive an equivalent volume of intrathecal saline co-administered with the spinal anesthetic. After surgery, bilateral ultrasound guided Quadratus Lumborum Block will be performed with 25 ml 0.5% Ropivacaine per side.
  Interventions: Procedure: Quadratus Lumborum Block; Drug: Intrathecal Saline
- Group 3 (Active Comparator): Group 3 will receive will receive intrathecal morphine with the spinal anesthetic. After the completion of surgery, bilateral ultrasound guided Quadratus Lumborum Block will be performed with 25 ml 0.5% Ropivacaine per side.
  Interventions: Procedure: Quadratus Lumborum Block; Drug: Intrathecal Morphine

INTERVENTIONS:
Procedure: Quadratus Lumborum Block — Quadratus Lumborum Block with Ropivacaine 0.5% will be done.
  Arms: Group 2; Group 3
Procedure: Sham Block — Sham block of Quadratus Lumborum will be done with Saline.
  Arms: Group 1
Drug: Intrathecal Morphine — Intrathecal Morphine 150 mcg will be co-administered with the spinal anesthetic.
  Other Names: Spinal Morphine
  Arms: Group 1; Group 3
Drug: Intrathecal Saline — Intrathecal Saline 0.15 mL will be co-administered with the spinal anesthetic.
  Other Names: Placebo
  Arms: Group 2

SUMMARY:
Most women having planned cesarean section receive spinal anesthetic for the procedure.

Typically, spinal opioids are administered during the same time as a component of multimodal analgesia to provide pain relief in the 16-24 hr period postoperatively. However, spinal opioids are frequently associated with adverse effects such as nausea, pruritus, sedation and occasionally respiratory depression.

The quadratus lumborum (QL) block is a regional analgesic technique which blocks T5-L1 nerve branches and has an evolving role in postoperative analgesia for lower abdominal surgeries and is a potential alternative to spinal opioids. There is some evidence that it may provide visceral along with somatic pain relief. It is a simple and safe technique that has been studied in lower abdominal surgeries, but has not been studied for pain relief after cesarean section.

If found effective, it will have the advantage of a reduction in opioid associated adverse effects while providing similar quality of analgesia. This block has evolved from the previously known transversus abdominis plane block.

We propose to undertake a study that will compare the relative efficacy of QL block with local anesthetic to spinal morphine. We will also study if it provides any incremental benefit when administered in addition to spinal morphine.

DETAILED DESCRIPTION:
This will be a randomized controlled double blinded trial.

Seventy five female patients belonging to American Society of Anesthesiologists status 1-3, age 18-45 yrs undergoing elective caesarean delivery will be included in this prospective study.

After obtaining informed consent, they will be randomized to one of the three groups by a computer-generated randomization. All patients will receive standard spinal anesthetic. They will be randomized to one of the three groups (n=25 per group).

Groups 1 and 3 will receive intrathecal morphine in addition to the spinal anesthestic. Group 2 will receive equal volume of saline added to the intrathecal mixture.

Ultrasound guided Quadratus Lumborum block will be done. Following negative aspiration, 25 mL of Ropivacaine 0.5% (Groups 2 and 3), or the same amount of saline (Group 1) will be injected in each side.

All patients will receive routine postoperative analgesia, including analgesics and oral morphine.

All patients will be assessed postoperatively by a blinded investigator at 6, 12 and 24h post-operatively.

ELIGIBILITY:
Inclusion Criteria:

* Elective cesarean delivery
* American Society of Anesthesiologists Physical Status 1-3
* Suitable for procedure to be carried out under spinal anesthesia

Exclusion Criteria:

* Inability to give informed consent or to co-operate with post-operative evaluation
* Allergy to local anesthetics, morphine, fentanyl, ropivacaine
* Ongoing major medical or psychiatric problems
* Chronic opioid use
* Major coagulopathy
* BMI>35 on first ante natal visit
* Pre-eclampsia
* Contraindication to neuraxial anesthesia

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2017-02-05 (Actual); Study Completion 2017-02-05 (Actual)

PRIMARY OUTCOMES:
Pain on movement at 12 hrs after surgery | 12 hours
  Numeric Rating Scale to evaluate pain scores at 12 h after surgery.

SECONDARY OUTCOMES:
Pain and Morphine consumption at 6,12 24 hrs after surgery. | 24 hours
  Numeric Rating Scale to evaluate pain scores.
Nausea at 6, 12, 24 hrs after surgery | 24 hours
  Nausea will be evaluated according to intensity. 0= no nausea; 1= nausea not requiring pharmacologic treatment; 2= nausea requiring pharmacologic treatment.
Chronic Wound Pain at 6 weeks | 6 weeks
  Development of chronic pain around incisional wound will be evaluated by phone interview.
Pruritus at 6, 12, 24 hrs after surgery | 24 hours
  Pruritus will be evaluated according to intensity 0= no pruritus; 1= pruritus not requiring pharmacologic treatment; 2= pruritus requiring pharmacologic treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Shalini Dhir, MD, FRCPC, Principal Investigator — University of Western Ontario, Canada
Locations (1):
- Victoria Hospital- LHSC, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided